CLINICAL TRIAL: NCT06278753
Title: Comparison of Standard Cystoscopy With Carbon Dioxide Cystoscopy Used to Evaluate Lower Urinary Tract Damage After Laparoscopic Hysterectomy.
Brief Title: Comparison of Standard Cystoscopy With Carbon Dioxide Cystoscopy
Status: Completed | Type: Observational
Sponsor: Tepecik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Abdurrahman Hamdi İnan, Associate Professor, Tepecik Training and Research Hospital
Other Study IDs: 2025/05/02
Record Dates: First submitted 2022-01-04; First posted 2024-02-26 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Bladder Injury; Ureter Injury; Surgical Injury; Complication of Surgical Procedure
Keywords: laparoscopic hysterectomy; lower urinary tract injury; cystoscopy
MeSH Terms: conditions — Intraoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard cystoscopy: Standard cystoscopy arm
- carbon dioxide cystoscopy: carbon dioxide cystoscopy arm
  Interventions: Diagnostic Test: carbon dioxide cystoscopy

INTERVENTIONS:
Diagnostic Test: carbon dioxide cystoscopy — Using carbon dioxide medium for filling bladder
  Groups: carbon dioxide cystoscopy

SUMMARY:
For the evaluation of the lower urinary tract after laparoscopic hysterectomy, routine standard saline cystoscopy and carbon dioxide cystoscopy will be compared.

DETAILED DESCRIPTION:
It was aimed to investigate whether routine cystoscopy with carbon dioxide is a safer and faster method for the evaluation of lower urinary tract injuries compared to standard saline cystoscopy. In addition, with this study, it will be studied whether bladder bleeding or intra-bladder masses can be evaluated more quickly and clearly.

ELIGIBILITY:
Inclusion Criteria:

1. laparoscopic hysterectomy for benign reasons planned patients
2. The operation will be performed in our hospital
3. Reporting preoperative endometrial and cervical samplings as benign
4. After discharge, control examinations will be carried out in our hospital.

Exclusion Criteria:

1. Abdominal, robotic or vaginal hysterectomies
2. malignant reporting of preoperative cervical and endometrial samplings
3. Patients do not want to participate in the study

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — cystoscopy after laparoscopic hysterectomy
Study Population: Patients who will undergo laparoscopic hysterectomy for benign reasons in our hospital
Sampling Method: Probability Sample
Enrollment: 540 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
It was aimed to evaluate the effectiveness and reliability of carbon dioxide cystoscopy. | one year

SECONDARY OUTCOMES:
It was aimed to evaluate the speed and image quality of carbon dioxide cystoscopy in detecting intravesical masses. | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Tepecik Training and Research Hospital, Izmir, Eurasia, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The data table will be shared with the researcher who requests it.